CLINICAL TRIAL: NCT03484689
Title: Mindfulness-based Cognitive Therapy (MBCT) for Type II Diabetes Mellitus (DM) Patients With High Diabetes Distress and Suboptimal DM Control: a Pilot Qusai-experimental Study
Brief Title: MBCT for DM Distress: a Pilot Qusai-experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Clinical assistant professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC17123
Record Dates: First submitted 2018-03-17; First posted 2018-04-02 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes-related distress; Mindfulness
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBCT arm (Other): 8-week MBCT program
  Interventions: Behavioral: Mindfulness-based cognitive therapy MBCT

INTERVENTIONS:
Behavioral: Mindfulness-based cognitive therapy MBCT — 8-week mindfulness-based cognitive therapy

SUMMARY:
Background: Diabetes-related distress (DRD) is very common among people with type II diabetes mellitus (DM). DRD led to poorer DM control and may led to adverse prognosis. Yet, there is no widely accepted or recommended DRD treatment.

Mindfulness was shown to relieve psychological distress in various physical and mental conditions.

Aim: as a pilot project, we aim to determine if mindfulness-based cognitive therapy (MBCT), which is one of the widely used mindfulness program, is feasible and acceptable and may improve DRD in our Chinese population.

Method: 20 Chinese participants with suboptimally controlled DM and high DRD will be recruited to a 8- week MBCT group. Pre-group and post-group (immediate and 2-month post-group) data including DRD score, quality-of life measures will be compared.

ELIGIBILITY:
Inclusion Criteria:

* received a clinical diagnosis of type II DM
* aged >=18
* can provide valid consent
* can speak Cantonese
* can read and write simple Chinese
* HbA1c >7%
* have CDDS score >=3

Exclusion Criteria:

* diagnosed active mental illness
* have severe hearing loss
* non-Chinese
* have active suicidal ideation as screened by Q9 of PHQ-9
* unwilling to join at least 6 out of 8 session of MBCT
* received mindfulness training in the past year or having regular mindfulness practice
* received psychotherapy last year
* severe physical illness limiting them from coming repeatedly to the group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-14 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of recruitment | From recruitment (1 April) till 20 patients are recruited (within 1 month)
  As a pilot study, we like to determine if it is feasible to recruit the target patients and measure the relevant outcomes. The number of patient approached and the number of patient recruited will be recorded
Dropout rate | Week 1 (start of MBCT, intervention) till week 8
  The proportion of patients attending at least 6 out of 8 classes

SECONDARY OUTCOMES:
Chinese Version of Diabetes Distress Scale (CDDS-15) | At pre-group (week1), immediate post-group (week8) and 2 months post-group (week16)
  A scale to diagnose and monitor Diabetes Related Distress. The scale ranged from score 0 to 6. The higher the score, the higher the distress.
9-item patient Health Questionnaire (PHQ-9) | At pre-group (week1), immediate post-group (week8) and 2 month post-group (week16)
  A scale of depression score. Higher scores signifies more severe depression. Possible score ranged from 0-27
The Audit of Diabetes-Dependent Quality of Life (ADDQOL) | At pre-group (week1), immediate post-group (week8) and 2 month post-group (week16)
  A measure of Diabetes specific quality of life. The possible score for each domain is from -9(most negative impact of diabetes) to +3 (most positive impact of diabetes). Domains include leisure work, journey, holiday, physical, family life, friendships and social life, personal relationship, sex life, physical appearance, self-confidence, motivation, reactions of other people, feelings about future, financial situation, living conditions, depend on others, freedom to eat, and freedom to drink. The total score is the weighted average of all the domain, so the total score also ranged from -9 to +3.

CONTACTS AND LOCATIONS:
Locations (1):
- Pok Oi Hopsital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Will be available only if requested by other investigators.